CLINICAL TRIAL: NCT07191938
Title: Comparison of Echo-guided Penile Block and Pudendal Block Under Neurostimulation for Perioperative Analgesia of Posthectomy in Pediatric Surgery: a Prospective, Randomized Study at Caen University Hospital
Brief Title: Posthectomy in Pediatric Elective Surgery : a Comparison of Perioperative Analgesia Using Echo-guided Penile Block and Pudendal Block With neurostimuLation Technique
Acronym: PinEAPPLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01470-47
Record Dates: First submitted 2025-07-02; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Care; Analgesia Assessment; Posthectomy; Postoperative Analgesia
Keywords: Neurostimulation guided pudendal block; US guided penile block; Security; Efficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided penile block (Experimental): The penile block is performed supine. After skin disinfection, the Buck's fascia is sonographically located, and the local anesthetic is injected close to the dorsal nerve of the penis in the plane after a negative aspiration test. The recommended dose is 0.1 ml/kg per side of ropivacaine 2 mg/ml. Injection is performed bilaterally. A subcutaneous injection of 1ml ropivacaine 2mg/ml is made at the base of the penis to ensure blockage of the perineal fibers.
  Interventions: Procedure: Ultrasound guided penile block
- Neurostimulation guided pudendal block (Active Comparator): The pudendal block is performed in the supine position, with the legs flexed. After skin disinfection and palpation of the ischial tuberosity, the neurostimulator needle, set at 0.5 mA, is inserted 1 cm medial to the tuberosity. Contraction of the anal sphincter enables the proximity of the pudendal nerve, originating from the S2, S3 and S4 nerve roots, to be identified. Once contraction has been obtained, local anaesthetic is injected using ropivacaine 2 mg/ml at a dose of 0.2 ml/kg per side, in the absence of blood reflux.
  Interventions: Procedure: Neurostimulation guided pudendal block

INTERVENTIONS:
Procedure: Ultrasound guided penile block — The penile block is performed supine. After skin disinfection, the Buck's fascia is sonographically located, and the local anesthetic is injected close to the dorsal nerve of the penis in the plane after a negative aspiration test (16). The recommended dose is 0.1 ml/kg per side of ropivacaine 2 mg/ml (8). Injection is performed bilaterally. A subcutaneous injection of 1ml ropivacaine 2mg/ml (i.e. 2mg) is made at the base of the penis to ensure blockage of the perineal fibers.
  Arms: Ultrasound guided penile block
Procedure: Neurostimulation guided pudendal block — The pudendal block is performed in the supine position, with the legs flexed. After skin disinfection and palpation of the ischial tuberosity, the neurostimulator needle, set at 0.5 mA, is inserted 1 cm medial to the tuberosity. Contraction of the anal sphincter enables the proximity of the pudendal nerve, originating from the S2, S3 and S4 roots, to be identified. Once contraction has been obtained, local anaesthetic is injected using ropivacaine 2 mg/ml at a dose of 0.2 ml/kg per side, in the absence of blood reflux.
  Arms: Neurostimulation guided pudendal block

SUMMARY:
Context : Posthectomy is a surgical procedure that concerns around 30% of the male population, mainly in pediatrics. As this procedure is mainly performed on an outpatient basis, the implementation of an enhanced rehabilitation protocol after surgery in pediatrics helps to reduce the incidence of postoperative pain, notably by providing multimodal analgesia, including locoregional anesthesia. Current recommendations from pediatric locoregional anesthesia societies favor penile block and the use of ultrasound in pediatric anesthesia to reduce anesthetic set-up time and the volume of local anesthetic, but also to increase the duration of sensory block and the success rate. However, several studies have shown the inferiority of penile block in anatomical landmarks compared with pudendal block under neurostimulation. As a result, pediatric anesthesiologists at Caen University Hospital prefer to use pudendal blocks under neurostimulation for posthectomy surgery. To date, no study has compared penile block under ultrasound with pudendal block under neurostimulation for postoperative analgesia after posthectomy surgery. On the other hand, a study of postoperative analgesia in hypospadias surgery showed a clear superiority of penile block under ultrasound over pudendal block in terms of both immediate postoperative pain and duration of postoperative analgesia. It therefore seems pertinent to compare these two techniques in posthectomy surgery.

Objective: We propose a prospective, open-label, non-inferiority study with the primary objective of comparing the efficacy of echo-guided penile block versus pudendal block in neurostimulation for posthectomy surgery.

Methods: This randomized, single-center study will include 240 patients divided into two groups. The experimental group will receive optimized medical and surgical management, with a penile block under ultrasound, while the control group will receive a pudendal block under neurostimulation. The planned duration of the study is 3 years.

Hypothesis tested: We hypothesize that ultrasound-guided penile block is non-inferior to neurostimulated pudendal block for postoperative analgesia in scheduled posthectomy surgery. The secondary objectives are to evaluate the time taken to perform the block, the volume of local anesthetic used, the need for sufentanil reinjection intraoperatively, the quantitative evaluation of analgesia using the EVENDOL score, the consumption of nalbuphine in the post anesthesia care unit, the occurrence of postoperative vomiting, and the length of stay in the post anesthesia care unit. The rate of complications related to the performance of locoregional anesthesia is also observed.

ELIGIBILITY:
Inclusion Criteria:

* All children aged over 3 months or 60 weeks post-conceptional age scheduled for outpatient posthectomy surgery

Exclusion Criteria:

* Recent airway infection.
* Contraindication to locoregional anesthesia: infection and/or loss of substance at the puncture site, congenital or acquired coagulopathy, product allergy.
* Contraindication to outpatient treatment: age < 12 weeks for healthy children or 60 weeks corrected age for premature babies, unbalanced pre-existing pathology (respiratory), ability to understand and comply with instructions (pre-operative fasting, taking painkillers at home and resumption of feeding), inability to ensure the presence of 2 adults including 1 parent on the return journey by car for children < 10 years old, easy access to care close to home.
* Emergency surgery.
* Coupled surgery (posthectomy + other surgery).
* Parents' refusal to participate in the study

Ages: 12 Weeks to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Failure of effective postoperative analgesia | Perioperative period : From anesthetic induction to discharge from the post- anesthesia care unit (12 hours maximum)
  It is defined by intense postoperative pain: an EVENDOL score ≥ 4 or the use of nalbuphine (0.1 to 0.2 mg/kg discontinuous) in the post anesthesia care unit "EVENDOL" is a French scale, which is an acronym of "EValuation ENfant DOuleur" or "Child pain assessment". This scale goes from 0 to 15, 0 is the absence of pain and 15 is the maximum pain. 4/15 is the threshold from which treatment is indicated.

SECONDARY OUTCOMES:
Locoregional anesthesia completion time | Peroperative period : From the end of skin disinfection to the removal of the locoregional anesthesia needle, assessed up to 30 minutes
  In seconds, defined as the time between the end of skin disinfection and removal of the locoregional anesthesia needle.
Volume of local anesthetic injected | Peroperative period : From skin disinfection to removal of the ALR needle, assessed up to 30 minutes
  Volume of local anesthetic injected (in mL/kg/side)
Intraoperative block failure rate | Peroperative period : From the beginning to the end of the surgery, assessed up to 2 hours
  Block failure is defined by the need to reinject sufentanil intraoperatively when systolic blood pressure or heart rate increases by more than 20% compared with the pre-incision heart rate, necessitating the consumption of intraoperative morphine.
Quantitative assessment of postoperative pain | Immediate post operative period : From the arrival to the discharge from the post anesthesia care unit, assessed up to 4 hours
  Quantitative assessment of postoperative pain using the EVENDOL score on arrival in the ICU, H+20 minutes, H+40 minutes and discharge from the post anesthesia care unit.
  As a reminder, EVENDOL" is a French scale, which is an acronym of "EValuation ENfant DOuleur" or "Child pain assessment". This scale goes from 0 to 15, 0 is the absence of pain and 15 is the maximum pain. 4/15 is the threshold from which treatment is indicated.
Nalbuphine consumption | Immediate postoperative period : From the arrival to the discharge from the post anesthesia care unit, assessed up to 4 hours
  Nalbuphine consumption in the post anesthesia care unit (in mg/kg)
Post operative vomiting | Immediate post operative period : From the arrival to the discharge from the post anesthesia care unit, assessed up to 4 hours
  Post operative vomiting and cosumption of ondansetron
Length of stay in post anesthesia care unit | Immediate postoperative period : From the arrival to the discharge from the post anesthesia care unit, assessed up to 4 hours
  In minutes
Adverse events related to local anesthesia | Perioperative period : From the completion of local anesthesia to the discharge from post anesthesia care unit, assessed up to 6 hours
  Signs of local anesthetic intoxication (neurological signs such as tinnitus, logorrhea or convulsion; tachycardia, hypotension), bleeding and hematoma at puncture site.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc Hanouz, MD, PhD, Study Chair — University Hospital, Caen
Locations (1):
- CHU de Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okoro C, Huang H, Cannon S, Low D, Liston DE, Richards MJ, Lendvay TS. The pudendal nerve block for ambulatory urology: What's old is new again. A quality improvement project. J Pediatr Urol. 2020 Oct;16(5):594.e1-594.e7. doi: 10.1016/j.jpurol.2020.07.025. Epub 2020 Jul 24. PMID 32819811
- [Background] Boisvert-Moreau F, Turcotte B, Albert N, Singbo N, Moore K, Boivin A. Randomized controlled trial (RCT) comparing ultrasound-guided pudendal nerve block with ultrasound-guided penile nerve block for analgesia during pediatric circumcision. Reg Anesth Pain Med. 2023 Mar;48(3):127-133. doi: 10.1136/rapm-2022-103785. Epub 2022 Nov 17. PMID 36396298
- [Background] Gnassingbe K, Akakpo-Numado KG, Anoukoum T, Kanassoua K, Kokoroko E, Tekou H. [The circumcision: why and how is it practiced in the newborn and the infant in the Lome teaching hospital?]. Prog Urol. 2009 Sep;19(8):572-5. doi: 10.1016/j.purol.2009.02.011. Epub 2009 Apr 3. French. PMID 19699456
- [Background] Aksu C, Akay MA, Sen MC, Gurkan Y. Ultrasound-guided dorsal penile nerve block vs neurostimulator-guided pudendal nerve block in children undergoing hypospadias surgery: A prospective, randomized, double-blinded trial. Paediatr Anaesth. 2019 Oct;29(10):1046-1052. doi: 10.1111/pan.13727. Epub 2019 Sep 2. PMID 31433895
- [Background] Pertek JP, Junke E, Coissard A, Vagner JC, Haberer JP. [Penile block in adults]. Ann Fr Anesth Reanim. 1992;11(1):82-7. doi: 10.1016/S0750-7658(05)80323-5. French. PMID 1443819
- [Background] Faraoni D, Gilbeau A, Lingier P, Barvais L, Engelman E, Hennart D. Does ultrasound guidance improve the efficacy of dorsal penile nerve block in children? Paediatr Anaesth. 2010 Oct;20(10):931-6. doi: 10.1111/j.1460-9592.2010.03405.x. PMID 20849498
- [Background] Tutuncu AC, Kendigelen P, Ashyyeralyeva G, Altintas F, Emre S, Ozcan R, Kaya G. Pudendal Nerve Block Versus Penile Nerve Block in Children Undergoing Circumcision. Urol J. 2018 May 3;15(3):109-115. doi: 10.22037/uj.v0i0.4292. PMID 29299888
- [Background] Naja Z, Al-Tannir MA, Faysal W, Daoud N, Ziade F, El-Rajab M. A comparison of pudendal block vs dorsal penile nerve block for circumcision in children: a randomised controlled trial. Anaesthesia. 2011 Sep;66(9):802-7. doi: 10.1111/j.1365-2044.2011.06753.x. Epub 2011 Jul 25. PMID 21790518
- [Background] Beydon L, Ecoffey C, Lienhart A, Puybasset L; Comite ICARE de Societe francaise d'anesthesie et de reanimation (Sfar). [Circumcision in children: an organizational or an ethical challenge?]. Ann Fr Anesth Reanim. 2012 May;31(5):442-6. doi: 10.1016/j.annfar.2012.01.038. Epub 2012 Mar 30. French. PMID 22464840

DOCUMENTS (1):
  • Informed Consent Form (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT07191938/ICF_000.pdf